CLINICAL TRIAL: NCT00316303
Title: The STIRR Intervention for Dually Diagnosed Clients
Brief Title: Effectiveness of the Screen, Test, Immunize, Reduce Risk, and Refer (STIRR) Intervention for People With Both a Mental and Substance Abuse Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH072556 (NIH); R01MH072556 (NIH); DAHBR 9A-ASNM
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Depression; Substance Abuse
Keywords: Serious Mental Illness; Dual Diagnosis; Mental Disorders; Substance-Related Disorders
MeSH Terms: conditions — HIV Infections; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depression; Substance-Related Disorders; Mental Disorders | interventions — twinrix

ARMS (2):
- 1 (Experimental): Participants will receive screening, testing, immunization, and risk reduction. Screening and testing will take place at study entry, immunization will occur at entry and after 3 and 6 months, and risk reduction will take place at study entry and after 3 and 6 months.
  Interventions: Drug: Twinrix
- 2 (Placebo Comparator): Participants will receive enhanced treatment as usual.
  Interventions: Behavioral: Enhanced treatment as usual

INTERVENTIONS:
Drug: Twinrix — This vaccine will be given in three parts: at entry and after 3 and 6 months.
  Arms: 1
Behavioral: Enhanced treatment as usual — Participants will receive comprehensive mental health services provided at each study site, education about blood-borne diseases, and referral to a local community health provider for blood testing, HAV and HBV immunizations, and any necessary treatments.
  Arms: 2

SUMMARY:
This study will determine the effectiveness of the STIRR (Screen, Test, Immunize, Reduce risk, and Refer) intervention in increasing rates of testing, immunization, referral, and treatment for blood-borne diseases, such as hepatitis and HIV, in people with both a mental disorder and a substance abuse disorder.

DETAILED DESCRIPTION:
People who have been dually diagnosed with a severe mental illness and a substance abuse disorder are at an elevated risk for contracting blood-borne infections, such as HIV, hepatitis B, and hepatitis C virus (HCV). Prevention, early detection, and treatment for these diseases are essential for this particular population. Research has shown that rates of HCV infection are 11 times higher in people with mental illnesses than in the general population. People with mental health illnesses and those with dual diagnoses should receive basic CDC-recommended services for risk screening and testing of HIV infection, AIDS, and hepatitis. They should also receive hepatitis A and B immunizations, risk reduction counseling, and referrals for medical care. However, most people with severe mental illnesses and substance abuse disorders do not receive the care they need. The STIRR (screen, test, immunize, reduce risk, and refer) intervention will provide necessary prevention and treatment services to an at-risk, under-treated population. This study will determine the effectiveness of the STIRR intervention in increasing rates of testing, immunization, referral, and treatment for blood-borne diseases, such as hepatitis and HIV, in people with both a mental disorder and a substance abuse disorder.

Participants in this open-label study will be recruited from two publicly funded community mental health agencies in Baltimore, MD. Participants will be randomly assigned to receive either enhanced treatment as usual or the STIRR intervention. Individuals assigned to STIRR will attend three sessions over the course of 6 months. The first session will involve education, personalized risk assessment, risk reduction counseling, pre-test counseling, blood testing, and an initial immunization with Twinrix for hepatitis A and B viruses (HAV and HBV). At the second session, participants will receive their test results, as well as post-test and risk reduction counseling, medical referral and linkage, if necessary, and a second Twinrix immunization. The third session will include an assessment of risk level and reinforcement of risk reduction, a final immunization, an assessment of progress on treatment and linkage, and behavior reinforcement or modification. Enhanced treatment as usual will entail comprehensive mental health services provided at each study site, education about blood-borne diseases, and referral to a local community health provider for blood testing, HAV and HBV immunizations, and any necessary treatments. All participants will be assessed for treatment outcomes at Month 6. A 12-month post-intervention follow-up will be carried out with the infected participants in the STIRR group to evaluate quality of care.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depression
* Diagnosis of a substance use disorder
* Enrolled in clinical care at Creative Alternatives or People Encouraging People for at least 3 months

Exclusion Criteria:

* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley D. Rosenberg, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Lisa Dixon, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Department of Psychaitry, Baltimore, Maryland, United States

REFERENCES:
- [Background] Rosenberg S, Brunette M, Oxman T, Marsh B, Dietrich A, Mueser K, Drake R, Torrey W, Vidaver R. The STIRR model of best practices for blood-borne diseases among clients with serious mental illness. Psychiatr Serv. 2004 Jun;55(6):660-4. doi: 10.1176/appi.ps.55.6.660. PMID 15175463
- [Background] Rosenberg SD, Drake RE, Brunette MF, Wolford GL, Marsh BJ. Hepatitis C virus and HIV co-infection in people with severe mental illness and substance use disorders. AIDS. 2005 Oct;19 Suppl 3:S26-33. doi: 10.1097/01.aids.0000192067.94033.aa. PMID 16251824
- [Derived] Rosenberg SD, Goldberg RW, Dixon LB, Wolford GL, Slade EP, Himelhoch S, Gallucci G, Potts W, Tapscott S, Welsh CJ. Assessing the STIRR model of best practices for blood-borne infections of clients with severe mental illness. Psychiatr Serv. 2010 Sep;61(9):885-91. doi: 10.1176/ps.2010.61.9.885. PMID 20810586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with co-occuring mental illness and substance use disorders who were receiving services from 2 publicly funded community mental health programs in Baltimore, MD.
Groups:
- STIRR Intervention: The STIRR Intervention involves Screening for HIV and hepatitis C risk factors, Testing for HIV and hepatitis B and C infection, Immunization against hepatitis A and B, and Reducing risk and Referring for medical treatment for persons testing positive for HIV and hepatitis C.
- Control Group: Participants will receive enhanced treatment as usual. This entails comprehensive mental health services provided at each study site, education about blood-borne diseases, and referral to a local community health provider for blood testing, hepatitis A (HAV) and hepatitis B (HBV)immunizations, and any necessary treatments.
Period: Overall Study
Arm/Group | STIRR Intervention | Control Group
Started | 118 | 118
Completed | 107 | 102
Not Completed | 11 | 16
Not completed — Lost to Follow-up | 11 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STIRR Intervention | Control Group | Total
Number analyzed (Participants) | 118 | 118 | 236
Age Continuous [Mean (Standard Deviation); unit: years] | 46.6 (8.5) | 46.3 (9.3) | 46.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 42 | 90
  Male | 70 | 76 | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 85 | 86 | 171
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 118 | 118 | 236

OUTCOME MEASURES:

1. Primary Outcome: Change in Immunization Status
Description: Of the participants that were not immunized at baseline, the number of participants who were immunized for Hepatitis A and B at 6 months.
Time Frame: Measured at 6 Months relative to Baseline
Measure: Number; unit: participants
Arm/Group | STIRR Intervention | Control Group
Number analyzed (Participants) | 96 | 86
participants | 73 | 4
Statistical Analysis 1: Comparison: STIRR Intervention vs Control Group; Test type: Superiority or Other; p < 0.001, Wald Chi-squared

2. Primary Outcome: Tested for Hepatitis C
Description: Participant self-report of being tested for hepatitis C
Time Frame: 6 Months
Measure: Number; unit: participants
Groups:
- STIRR Intervention: The STIRR Intervention involved Screening for HIV and hepatitis C risk factors, Testing for HIV and hepatitis B and C infection, Immunization against hepatitis A and B, and Reducing risk and Referring for medical treatment for persons testing positive for HIV and hepatitis C.
- Control Group: Participants will receive enhanced treatment as usual. This entails comprehensive mental health services provided at each study site, education about blood-borne diseases, and referral to a local community health provider for blood testing, hepatitis A and hepatitis B immunizations, and any necessary treatments.
Arm/Group | STIRR Intervention | Control Group
Number analyzed (Participants) | 81 | 69
participants | 70 | 10
Statistical Analysis 1: Comparison: STIRR Intervention vs Control Group; Test type: Superiority or Other; p < 0.001, Wald Chi-squared

3. Primary Outcome: Tested for Hepatitis B
Description: Participant self-report of being tested for hepatitis B
Time Frame: 6 Months
Measure: Number; unit: participants
Groups:
- Control Group: Participants will receive enhanced treatment as usual. This entails comprehensive mental health services provided at each study site, education about blood-borne diseases, and referral to a local community health provider for blood testing, HAV and HBV immunizations, and any necessary treatments.
Arm/Group | STIRR Intervention | Control Group
Number analyzed (Participants) | 80 | 73
participants | 69 | 14
Statistical Analysis 1: Comparison: STIRR Intervention vs Control Group; Test type: Superiority or Other; p < 0.001, Wald Chi-squared

4. Primary Outcome: Tested for HIV
Description: Participant self-report of being tested for HIV
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | STIRR Intervention | Control Group
Number analyzed (Participants) | 21 | 13
participants | 18 | 6
Statistical Analysis 1: Comparison: STIRR Intervention vs Control Group; Test type: Superiority or Other; p = 0.011, Wald Chi-squared

5. Primary Outcome: Referral for Medical Care
Description: For participants infected with hepatitis C, their self-report of being referred for medical care.
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | STIRR Intervention | Control Group
Number analyzed (Participants) | 21 | 16
participants | 17 | 12
Statistical Analysis 1: Comparison: STIRR Intervention vs Control Group; Test type: Superiority or Other; p = 0.6, Chi-squared

ADVERSE EVENTS:
Arm/Group | STIRR Intervention | Control Group
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/118
Other Adverse Events (participants affected / at risk) | 0/118 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes